CLINICAL TRIAL: NCT00400179
Title: An Open-Label Multicenter, Randomized, Phase 3 Study of S-1 in Combination With Cisplatin Against 5-Fu in Combination W/ Cisplatin in Patients W/ Advanced Gastric Cancer Previously Untreated W/ Chemotherapy for Advanced Disease
Brief Title: A Safety and Efficacy Study in Patients With Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPU S-1301; NCT00128609 (obsolete NCT alias)
Record Dates: First submitted 2005-06-30; First posted 2006-11-16 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S-1 plus cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): In Arm A, S-1 25 mg/m² was administered orally BID from Day 1 through Day 21 followed by a recovery period from Days 22 through Day 28. On Day 1, the morning dose of S-1 was administered before cisplatin 75 mg/m2 administration as a 1- to 3-hour IV infusion. This regimen was repeated every 4 weeks. S-1 was administered one hour before or one hour after a meal with a glass of water (approximately 100 mL).
  Interventions: Drug: S-1/Cisplatin
- B (Active Comparator): In Arm B, 5-FU 1000 mg/m2/24 hours was administered by continuous intravenous infusion (CIV) over 120 hours (on Days 1 through 5). This regimen was repeated every 4 weeks. 5-FU CIV followed cisplatin infusion on Day 1. All 5-FU used in this study was commercially available product.
  Interventions: Drug: 5-FU/cisplatin

INTERVENTIONS:
Drug: S-1/Cisplatin — In Arm A, S-1 25 mg/m2 was taken orally two times daily for 21 days followed by a 7-day recovery period. The patient was instructed to have nothing by mouth (NPO 1 hour prior to and 1 hour after S-1 administration. S-1 was taken with approximately 8 ounces of water and prior to cisplatin infusion on Day 1.
  Cisplatin 75 mg/m2 was administered as a 1- to 3-hour IV infusion after the morning dose of S-1 on Day 1 of each cycle. This regimen was repeated every 4 weeks with a maximum of 6 cycles of treatment for cisplatin.
  Arms: A
Drug: 5-FU/cisplatin — In Arm B, 5-FU 1000 mg/m2/24 hours was administered CIV on Days 1 through 5 following cisplatin 100 mg/m2 administered IV as a 1- to 3-hour infusion on Day 1. This regimen was repeated every 4 weeks with a maximum of 6 cycles of treatment for cisplatin.
  Arms: B

SUMMARY:
This is an open-label, international, two-arm, parallel, randomized, Phase 3 study evaluating the efficacy and safety of S-1/cisplatin versus 5-FU/cisplatin in patients with advanced gastric cancer previously untreated with chemotherapy for advanced disease. Patients will be randomly assigned (1:1) to S-1/cisplatin (experimental arm) or 5-FU/cisplatin (control arm). Patients will be stratified by number of metastatic sites (one vs. more than one), locally advanced or metastatic disease, prior adjuvant therapy (yes or no), measurable or non-measurable disease, and center.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study:

* Has given written informed consent
* Has histologically confirmed, unresectable, locally advanced (Stage IV) or metastatic gastric cancer, including adenocarcinoma of the gastro-esophageal junction
* Has measurable or evaluable but non-measurable disease, defined as follows:

  * Measurable Disease - Patients with measurable disease as defined by RECIST criteria, i.e., the presence of at least one measurable lesion. A measurable lesion is one that can be accurately measured in at least one dimension with the longest diameter >_ 20 mm using conventional techniques or >_ 10 mm using spiral Computed Tomography (CT)scan. Locally recurrent disease (other than primary) is accepted if there is at least one measurable lesion (i.e. peritoneal mass, lymph node, etc.)
  * Evaluable but Non-measurable Disease - Patients with all lesions below the limits defined above for measureable disease (i.e., longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT) excluding those patients with only a primary lesion and/or with only non-evaluable cancer such as bone metastases, ascites, pleural or pericardia effusions, lymphangitic carcinomatosis of the skin or lung, previously irradiated lesions not in progression, or peritoneal carcinomatosis < 10 mm in diameter with conventional imaging techniques.
* No prior palliative chemotherapy is permitted. Adjuvant and /or neo-adjuvant chemotherapy is permitted if more than 12 months have elapsed between the end of adjuvant or neo-adjuvant therapy and first recurrence. This does not qualify as 1st line therapy.
* Is able to take medications orally
* Is >_ 18 years of age
* Is at least 3 weeks from prior major surgery
* Is at least 4 weeks from prior radiotherapy
* Has a ECOG performance status 0 to 1
* Has adequate organ function as defined by the following criteria:

  * AST (SGOT) and ALT (SGPT) <_ 2.5 x ULN; if liver function abnormalities are due to underlying liver metastasis, AST (SGOT) and ALT (SGPT) <_ 5 x ULN
  * Total serum bilirubin of <_ 1.5 x ULN
  * Absolute granulocyte count of >_ 1,500/mm (i.e. >_ 1.5 x 10/L by International Units (IU)
  * Platelet count >_ 100,000/mm (IU: >_ 100 x 10/L
  * Hemoglobin value of >_ 9.0 g/dL
  * Calculated creatinine clearance >_ 60 mL/min (Cockcroft-Gault formula)
* Is willing and able to comply with scheduled visits, treatment plans, laboratory tests and other study procedures

Exclusion Criteria:

Exclude a patient from this study if he/she does not fulfill the inclusion criteria, or if any of the following conditions are observed:

* Has had a treatment with any of the following within the specified timeframe prior to study drug administration:

  * Any prior palliative chemotherapy or any previous therapy for malignancy, including any chemotherapy, immunotherapy, biologic or hormonal therapy, within the past 5 years.
  * Adjuvant or neo-adjuvant therapy within the past 12 months
  * Concurrent treatment with any investigational anti-cancer agent
  * Prior cisplatin as neo-adjuvant and /or adjuvant chemotherapy with cumulative dose > 300 mg/m
  * > 25% of marrow-bearing bone radiated
  * Concurrent treatment with an investigational agent or within 30 days from randomization
  * Concurrent enrollment in another clinical study
* Has a serious illness or medical condition(s) including, but not limited to the following:

  * Known brain or leptomeningeal metastases
  * Uncontrolled ascites requiring drainage at least twice a week
  * Other malignancies within the past 5 years, except adequately treated carcinoma-in-situ of the cervix or non-melanoma skin cancer
  * Myocardial infarction within the last 6 months, severe/unstable angina, congestive heart failure New York Heart Association (NYHA) class III or IV
  * Chronic nausea, vomiting or diarrhea
  * Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS-related illness
  * Psychiatric disorder that may interfere with consent and/or protocol compliance
  * Known neuropathy, Grade 2 or higher
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgement of the Investigator would make the patient inappropriate for entry into this study
* Is receiving concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:

  * Sorivudine, uracil, cimetidine, folinic acid, and dipyridamole (may enhance S-1 activity)
  * Allopurinol (may diminish S-1 activity
  * Phenytoin (S-1 may enhance phenytoin activity)
  * Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 activity)
* Is receiving concomitant treatment with drugs interacting with 5-FU:

  * Sorivudine, uracil, cimetidine, folinic acid, and dipyridamole(may enhance 5-FU activity)
  * Allopurinol (may diminish 5-FU activity)
  * Phenytoin (5-FU may enhance phenytoin activity)
* Is receiving concomitant treatment with drugs interacting with cisplatin:

  * Phenytoin (cisplatin may diminish phenytoin activity)
  * Aminoglycosides (should be avoided within 8 days after cisplatin administration)
  * Ethyol (may diminish cisplatin activity
* Is a pregnant or lactating female
* Has known hypersensitivity to 5-FU or cisplatin
* Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Benedetti, MD, Study Director — Taiho Oncology, Inc.
Locations (33):
- United States (32):
  - Clearview Cancer Center, Huntsville, Alabama
  - Saint Joseph Medical Center, Burbank, California
  - Dr. Ronald Yanagihara, Gilroy, California
  - Norris Cancer Center, Los Angeles, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Saint Francis Memorial Hospital, San Francisco, California
  - Premiere Oncology, Santa Monica, California
  - Western Hematology/Oncology, Lakewood, Colorado
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Alexandar Rosemurgy, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Oncology and Hematology, Metairie, Louisiana
  - St. Lukes Cancer Care Center, Duluth, Minnesota
  - Neuroscience Center, St Louis, Missouri
  - St. Louis University Cancer Center, St Louis, Missouri
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - AHS Lovelace Medical Group,LLC, Albuquerque, New Mexico
  - New Mexico Cancer Center Associates, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Hoo Chun, MD, Hawthorne, New York
  - Hematology/Oncology Associates of Rockland, New City, New York
  - New Bern Cancer Care, New Bern, North Carolina
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - Lexington Oncology Associates, Chattanooga, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- CHUM Hopital Saint-Luc, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bodoky G, Scheulen ME, Rivera F, Jassem J, Carrato A, Moiseyenko V, Vynnychenko I, Prausova J, Van Laethem JL, Cascinu S, Ajani JA. Clinical Benefit and Health-Related Quality of Life Assessment in Patients Treated with Cisplatin/S-1 Versus Cisplatin/5-FU: Secondary End Point Results From the First-Line Advanced Gastric Cancer Study (FLAGS). J Gastrointest Cancer. 2015 Jun;46(2):109-17. doi: 10.1007/s12029-014-9680-1. PMID 25707610
- [Derived] Ajani JA, Buyse M, Lichinitser M, Gorbunova V, Bodoky G, Douillard JY, Cascinu S, Heinemann V, Zaucha R, Carrato A, Ferry D, Moiseyenko V. Combination of cisplatin/S-1 in the treatment of patients with advanced gastric or gastroesophageal adenocarcinoma: Results of noninferiority and safety analyses compared with cisplatin/5-fluorouracil in the First-Line Advanced Gastric Cancer Study. Eur J Cancer. 2013 Nov;49(17):3616-24. doi: 10.1016/j.ejca.2013.07.003. Epub 2013 Jul 27. PMID 23899532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted between May 18, 2005 and March 7, 2008 in 24 countries including the United States. Study centers were also located in Canada, Eastern and Western Europe, South America, Australia, and ex-Soviet Union block of nations.
Groups:
- S-1/Cisplatin: In the S-1/cisplatin arm, S-1 25 mg/m2 was taken orally two times daily for 21 days followed by a 7-day recovery period. The patient was instructed to have nothing by mouth 1 hour prior to and 1 hour after S-1 administration. S-1 was taken with a glass of water and prior to cisplatin infusion on Day 1.
  Cisplatin 75 mg/m2 was administered as a 1- to 3-hour intravenous (IV) infusion after the morning dose of S-1 on Day 1 of each cycle. This regimen was repeated every 4 weeks with a maximum of 6 cycles of treatment.
- 5-FU/Cisplatin: In the 5-FU/cisplatin arm, 5-FU 1000 mg/m2/24 hours was administered by continuous intravenous infusion on Days 1 through 5 following cisplatin 100 mg/m2 administered IV as a 1- to 3-hour infusion on Day 1. This regimen was repeated every 4 weeks with a maximum of 6 cycles.
Period: Overall Study
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin
Started | 527 (Signed informed consent form and randomized) | 526
Completed | 521 (Received Treatment) | 508
Not Completed | 6 | 18
Not completed — Adverse Event | 2 | 2
Not completed — Death | 1 | 2
Not completed — Withdrew Consent | 1 | 5
Not completed — Disease progression | 1 | 1
Not completed — Intercurrent illness | 0 | 1
Not completed — Investigator judgment | 0 | 1
Not completed — Randomization error/patient ineligible | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin | Total
Number analyzed (Participants) | 521 | 508 | 1029
Age, Continuous [Median (Full Range); unit: Years]
  Baseline Measure Data (descriptive stats, median) | 59.0 [18 to 83] | 59.0 [18 to 85] | 59.0 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 161 | 300
  Male | 382 | 347 | 729
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 6 | 10
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 447 | 438 | 885
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 61 | 53 | 114
Body surface area (BSA) Categories [Number; unit: Participants]
  </=1.29 m2 | 4 | 5 | 9
  1.30-1.49 m2 | 46 | 44 | 90
  1.50-1.69 m2 | 118 | 147 | 265
  1.70-1.89 m2 | 208 | 181 | 389
  1.90-2.09 m2 | 114 | 93 | 207
  2.10-2.29 m2 | 29 | 34 | 63
  >/=2.30 m2 | 2 | 4 | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — 0=Fully active, able to carry on all pre-disease performance without restriction
  1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 226 | 200 | 426
    1 | 295 | 308 | 603
Tissue Type [Number; unit: Participants] — Patients can have more than one tissue type and are included under each type.
  Participants
    Papillary adenocarcinoma | 15 | 15 | 30
    Tubular adenocarcinoma | 132 | 113 | 245
    Well-differentiated | 20 | 17 | 37
    Moderately-differentiated | 105 | 91 | 196
    Unknown | 7 | 5 | 12
    Poorly differentiated adenocarcinoma | 210 | 189 | 399
    Signet-ring cell carcinoma | 75 | 95 | 170
    Mucinous adenocarcinoma | 28 | 32 | 60
    Other | 97 | 94 | 191
    Adenocarcinoma NOS | 87 | 87 | 174
    Poorly differentiated cancer | 7 | 2 | 9
    Unknown/not specified | 1 | 1 | 2
    Other types | 2 | 4 | 6
Anatomical Location of Primary Lesion [Number; unit: Participants]
  Stomach | 438 | 417 | 855
  Gastroesophageal junction | 82 | 88 | 170
  Stomach and gastroesophageal junction | 1 | 3 | 4
Extent of Disease [Number; unit: Participants]
  Locally advanced | 23 | 20 | 43
  1 metastatic site | 157 | 161 | 318
  >/=2 metastatic sites | 340 | 327 | 667
  Not assessed | 1 | 0 | 1
Disease Measurability [Number; unit: Participants]
  Measureable disease | 499 | 485 | 984
  Non-measurable disease | 21 | 22 | 43
  Nonevaluable disease | 0 | 1 | 1
  No disease present | 1 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Overall Response Rate (ORR)
Description: The proportion of patients with objective evidence of complete response (CR) or partial response (PR) based on tumor response assessments. Per the Response Evaluation Criteria in Solid tumors (RECIST), CR was defined as the disappearance of all target lesions for at least 4 weeks, and PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Data cutoff was 07 March 2008 (12 months after last patient randomized).
Measure: Number (95% Confidence Interval); unit: Percentage of patients in each group
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin
Number analyzed (Participants) | 402 | 385
Percentage of patients in each group | 29.1 [24.7 to 33.8] | 31.9 [27.3 to 36.9]
Statistical Analysis 1: Comparison: S-1/Cisplatin vs 5-FU/Cisplatin; Test type: Superiority or Other; p = 0.3952, Fisher Exact

2. Secondary Outcome: Duration of Response (DR)
Description: Duration of response was defined as the time from date of first confirmed response (CR or PR) to date of first progressive disease (PD) or death. Per the RECIST criteria, definitions were as follows: CR was the disappearance of all target lesions for at least 4 weeks, PR was at least a 30% decrease in the sum of the longest diameter of target lesions, and PD was at least a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Data cutoff was 07 March 2008 (12 months after last patient was randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin
Number analyzed (Participants) | 402 | 385
Months | 6.5 [5.8 to 7.4] | 5.8 [5.5 to 6.1]
Statistical Analysis 1: Comparison: S-1/Cisplatin vs 5-FU/Cisplatin; Test type: Superiority or Other; p = 0.0808, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.57 to 1.03]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The time from randomization to date of first documented PD or date of death, whichever occurred first.
Time Frame: From date of randomization until date of first documented PD, date of death, or until data cutoff on 07 March 2008 (12 months after last patient randomized), whichever came first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin
Number analyzed (Participants) | 521 | 508
Months | 4.8 [4.0 to 5.5] | 5.5 [4.4 to 5.8]
Statistical Analysis 1: Comparison: S-1/Cisplatin vs 5-FU/Cisplatin; Test type: Superiority or Other; p = 0.9158, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.14]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: The time from randomization to date of permanent discontinuation of S-1 or 5-FU, first documented PD, or death, whichever occurred first.
Time Frame: From date of randomization until date of permanent discontinuation of S-1 or 5-FU, first documented PD, death, or data cutoff on 07 March 2008 (12 months after last patient randomized), whichever came first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin
Number analyzed (Participants) | 521 | 508
Months | 3.8 [3.7 to 4.0] | 3.8 [3.7 to 4.4]
Statistical Analysis 1: Comparison: S-1/Cisplatin vs 5-FU/Cisplatin; Test type: Superiority or Other; p = 0.0320, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.77 to 0.99]

5. Primary Outcome: Median Survival
Description: Survival was defined as the time from the date of randomization to the time of death (from any cause) for each patient.
Time Frame: The cutoff date for survival analysis was 07 March 2008 (12 months after last patient randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin
Number analyzed (Participants) | 521 | 508
Months | 8.6 [7.9 to 9.5] | 7.9 [7.2 to 8.5]
Statistical Analysis 1: Comparison: S-1/Cisplatin vs 5-FU/Cisplatin; Test type: Superiority or Other; p = 0.1983, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.80 to 1.05]

ADVERSE EVENTS:
Time Frame: From the start of study drug administration until 12 months after last patient randomized
Arm/Group | S-1/Cisplatin | 5-FU/Cisplatin
Serious Adverse Events (participants affected / at risk) | 257/521 | 248/508
Other Adverse Events (participants affected / at risk) | 514/521 | 504/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-1/Cisplatin (N=521) | 5-FU/Cisplatin (N=508)
Anaemia (Blood and lymphatic system disorders) | 33 (37) | 31 (38)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 31 (34)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 31 (34)
Pancytopenia (Blood and lymphatic system disorders) | 2 (5) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (11) | 17 (18)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal haemorrhage (Endocrine disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Vitreious floaters (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 13 (13)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 5 (5) | 4 (4)
Gastric perforation (Gastrointestinal disorders) | 4 (4) | 4 (4)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (13) | 8 (8)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 5 (6) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 3 (3)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (18) | 10 (13)
Obstruction gastric (Gastrointestinal disorders) | 6 (6) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 3 (4)
Periproctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Prepyloric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 24 (30)
Subileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 23 (23) | 17 (21)
Asthenia (General disorders) | 4 (4) | 4 (4)
Catheter site pain (General disorders) | 0 (0) | 2 (2)
Catheter thrombosis (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 9 (9) | 1 (1)
Disease progression (General disorders) | 53 (53) | 34 (34)
Fatigue (General disorders) | 8 (10) | 6 (7)
Generalised Oedema (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 10 (11)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 10 (10) | 1 (1)
Sudden death (General disorders) | 2 (2) | 3 (3)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (5) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Broncopneumonia (Infections and infestations) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 4 (4)
Catheter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Central line infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 1 (1)
Genital candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Neutropenic sepsis (Infections and infestations) | 3 (3) | 5 (5)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyothorax (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 3 (3)
Septic shock (Infections and infestations) | 3 (3) | 10 (10)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device migration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 4 (4)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Urine electrolytes increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (8) | 2 (2)
Cachexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 21 (21) | 32 (41)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 8 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 6 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (9) | 3 (4)
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acoustic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 3 (4)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 5 (6) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 3 (3) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 5 (5) | 9 (9)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 11 (11)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal tubular disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 2 (2) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 17 (18)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 3 (4)
Hypovolaemic shock (Vascular disorders) | 4 (4) | 1 (1)
Iliac artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Pelvis venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-1/Cisplatin (N=521) | 5-FU/Cisplatin (N=508)
Anaemia (Blood and lymphatic system disorders) | 229 (404) | 234 (380)
Neutropenia (Blood and lymphatic system disorders) | 149 (383) | 240 (588)
Thrombocytopenia (Blood and lymphatic system disorders) | 92 (174) | 116 (190)
Leukopenia (Blood and lymphatic system disorders) | 91 (224) | 117 (254)
Lymphopenia (Blood and lymphatic system disorders) | 26 (54) | 34 (126)
Granulocytopenia (Blood and lymphatic system disorders) | 18 (60) | 10 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10) | 35 (38)
Leukocytosis (Blood and lymphatic system disorders) | 8 (13) | 15 (22)
Tinnitus (Ear and labyrinth disorders) | 29 (76) | 44 (75)
Deafness (Ear and labyrinth disorders) | 11 (12) | 24 (27)
Lacrimation increased (Eye disorders) | 32 (62) | 6 (8)
Vision blurred (Eye disorders) | 18 (81) | 9 (13)
Nausea (Gastrointestinal disorders) | 321 (778) | 342 (913)
Vomiting (Gastrointestinal disorders) | 260 (616) | 281 (693)
Diarrhoea (Gastrointestinal disorders) | 152 (329) | 195 (331)
Abdominal pain (Gastrointestinal disorders) | 131 (219) | 114 (205)
Constipation (Gastrointestinal disorders) | 120 (296) | 133 (219)
Abdominal pain upper (Gastrointestinal disorders) | 66 (125) | 67 (85)
Dyspepsia (Gastrointestinal disorders) | 46 (86) | 30 (41)
Stomatitis (Gastrointestinal disorders) | 33 (74) | 153 (321)
Flatulence (Gastrointestinal disorders) | 31 (49) | 10 (11)
Dysphagia (Gastrointestinal disorders) | 26 (29) | 42 (54)
Ascites (Gastrointestinal disorders) | 25 (27) | 13 (15)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 19 (19) | 14 (15)
Abdominal distension (Gastrointestinal disorders) | 16 (23) | 18 (20)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 (21) | 8 (9)
Fatigue (General disorders) | 205 (505) | 200 (329)
Asthenia (General disorders) | 88 (124) | 96 (152)
Pyrexia (General disorders) | 72 (112) | 61 (80)
Disease progression (General disorders) | 55 (55) | 35 (35)
Oedema peripheral (General disorders) | 53 (81) | 46 (56)
Performance status decreased (General disorders) | 35 (36) | 42 (49)
Chest pain (General disorders) | 27 (38) | 23 (30)
Mucosal inflammation (General disorders) | 20 (27) | 152 (330)
Chills (General disorders) | 16 (20) | 10 (13)
Injection site reaction (General disorders) | 5 (11) | 15 (21)
Hyperbilirubinaemia (Hepatobiliary disorders) | 32 (47) | 15 (21)
Nasopharyngitis (Infections and infestations) | 16 (19) | 9 (9)
Oral candidiasis (Infections and infestations) | 3 (3) | 22 (31)
Weight decreased (Investigations) | 148 (157) | 164 (173)
Creatinine renal clearance decreased (Investigations) | 37 (43) | 61 (72)
Blood creatinine increased (Investigations) | 35 (45) | 62 (78)
Haemoglobin decreased (Investigations) | 26 (35) | 22 (31)
Aspartate aminotransferase increased (Investigations) | 25 (29) | 18 (25)
Blood alkaline phosphatase increased (Investigations) | 23 (25) | 28 (32)
Neutrophil count decreased (Investigations) | 22 (41) | 29 (61)
Alanine aminotransferase increased (Investigations) | 16 (18) | 19 (25)
Blood LDH increased (Investigations) | 16 (22) | 19 (24)
Blood urea increased (Investigations) | 15 (28) | 30 (35)
Platelet count decreased (Investigations) | 15 (28) | 27 (46)
White blood cell count decreased (Investigations) | 14 (22) | 24 (44)
Glomerular filtration rate decreased (Investigations) | 6 (6) | 15 (18)
Anorexia (Metabolism and nutrition disorders) | 164 (306) | 177 (310)
Dehydration (Metabolism and nutrition disorders) | 63 (81) | 79 (114)
Hypomagnesaemia (Metabolism and nutrition disorders) | 52 (91) | 52 (74)
Hyponatraemia (Metabolism and nutrition disorders) | 38 (55) | 41 (51)
Hypokalaemia (Metabolism and nutrition disorders) | 36 (52) | 85 (133)
Decreased appetite (Metabolism and nutrition disorders) | 26 (31) | 30 (62)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26 (36) | 46 (63)
Hypocalcaemia (Metabolism and nutrition disorders) | 23 (26) | 36 (45)
Hyperglycaemia (Metabolism and nutrition disorders) | 19 (28) | 21 (32)
Hyperkalaemia (Metabolism and nutrition disorders) | 17 (18) | 19 (20)
Hypophosphataemia (Metabolism and nutrition disorders) | 10 (12) | 30 (43)
Back pain (Musculoskeletal and connective tissue disorders) | 45 (58) | 44 (57)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (29) | 19 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (31) | 8 (11)
Dizziness (Nervous system disorders) | 53 (128) | 36 (72)
Headache (Nervous system disorders) | 50 (127) | 51 (72)
Dysgeusia (Nervous system disorders) | 48 (128) | 50 (79)
Peripheral sensory neuropathy (Nervous system disorders) | 42 (80) | 44 (59)
Paraesthesia (Nervous system disorders) | 18 (23) | 21 (29)
Neuropathy peripheral (Nervous system disorders) | 14 (18) | 33 (35)
Insomnia (Psychiatric disorders) | 40 (173) | 67 (129)
Depression (Psychiatric disorders) | 14 (16) | 17 (17)
Anxiety (Psychiatric disorders) | 10 (11) | 31 (39)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 37 (98) | 45 (99)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (37) | 36 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (89) | 33 (46)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 15 (20)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 15 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 31 (50) | 104 (111)
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 28 (52) | 13 (27)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 27 (29) | 17 (21)
Rash (Skin and subcutaneous tissue disorders) | 27 (53) | 21 (29)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 20 (62) | 13 (22)
Hypotension (Vascular disorders) | 24 (26) | 24 (27)
Hypertension (Vascular disorders) | 21 (31) | 20 (25)
Deep vein thrombosis (Vascular disorders) | 14 (14) | 22 (24)
Phlebitis (Vascular disorders) | 8 (10) | 23 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Taiho agreements vary with individual investigators, but do not prohibit any from publishing. Taiho is provided time to review material discussing trial results (generally 30 to 120 days with possible extension), and can remove undisclosed confidential, proprietary and intellectual property rights-related information. Authors have final control and approval of publication content of final study results. The investigator agrees not to publish any results before the first multicenter publication.